CLINICAL TRIAL: NCT02144012
Title: A Randomized, Multicenter, Open-Label Phase III Study to Evaluate the Efficacy and Safety of Trastuzumab Emtansine Versus the Combination of Trastuzumab Plus Docetaxel as First-Line Treatment of Patients With Her2-Positive Progressive Or Recurrent Locally Advanced Or Metastatic Breast Cancer.
Brief Title: A Study to Evaluate the Efficacy and Safety of Trastuzumab Emtansine Versus the Combination of Trastuzumab Plus Docetaxel in Patients With HER2-positive Breast Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YO28405
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Ado-Trastuzumab Emtansine; Docetaxel

ARMS (2):
- Arm A: Trastuzumab emtansine (Experimental): Participants will be administered trastuzumab emtansine once every three weeks (Q3W). Participants may remain on study treatment until investigator assessed disease progression, unacceptable toxicity, or Sponsor study termination occurs, whichever occurs first.
  Interventions: Drug: Trastuzumab Emtansine
- Arm B: Trastuzumab + Docetaxel (Active Comparator): Participants will be administered trastuzumab plus docetaxel Q3W. Participants may remain on study treatment until investigator assessed disease progression, unacceptable toxicity, or Sponsor study termination occurs, whichever occurs first.
  Interventions: Drug: Trastuzumab; Drug: Docetaxel

INTERVENTIONS:
Drug: Trastuzumab — For the first three-week cycle, trastuzumab was administered IV at 8 mg/kg. For subsequent cycles, trastuzumab was administered IV at 6 mg/kg Q3W.
  Other Names: Herceptin
  Arms: Arm B: Trastuzumab + Docetaxel
Drug: Trastuzumab Emtansine — Trastuzumab emtansine 3.6 milligrams/kilogram (mg/kg) was administered intravenously (IV) over 30-90 minutes Q3W.
  Other Names: Kadcyla
  Arms: Arm A: Trastuzumab emtansine
Drug: Docetaxel — Docetaxel was administered IV at either 75 milligrams/square meter (mg/m^2) or 100 mg/m^2 Q3W.
  Arms: Arm B: Trastuzumab + Docetaxel

SUMMARY:
This is a Phase III, randomized, multicenter, multinational, two-arm, open-label clinical trial to investigate a first-line treatment of participants with human epidermal growth factor receptor-2 (HER2)-positive metastatic breast cancer. The study will enroll patients with HER2-positive, unresectable, locally advanced breast cancer (BC) if they have recurrent disease or progressive disease (PD) despite primary multi-modality therapy, and/or metastatic BC if they have not received prior chemotherapy for their metastatic disease. Eligible participants at up to approximately 40 sites in the Asia-Pacific region will be randomized in a 2:1 ratio to receive trastuzumab emtansine (Arm A) or trastuzumab plus docetaxel (Arm B). All study drugs will be administered at in-clinic visits occurring every three weeks during the treatment phase. Trastuzumab plus docetaxel was chosen as the comparator in the control group (Arm B), as it represents a common first-line treatment option used in this patient population in China and other Asia-Pacific countries.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* HER2-positive disease, as defined by an immunohistochemistry test score of 3+ and/or in situ hybridization positivity, prospectively confirmed by a Sponsor-designated central laboratory prior to enrollment
* Histologically or cytologically confirmed adenocarcinoma of the breast with locally recurrent or metastatic disease appropriate for chemotherapy
* Patients must have measurable and/or non-measurable disease that is evaluable per the Response Evaluation Criteria in Solid Tumors (RECIST) criteria, version 1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate organ function
* For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use two adequate non-hormonal forms of contraception during treatment and for at least 6 months after the last dose of study drug

Exclusion Criteria:

* Pregnancy or lactation
* Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease; wound healing disorders; ulcers; bone fractures, except bone fractures because of disease under study)
* Currently known active infection with HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV)
* Major surgical procedure or significant traumatic injury within approximately 28 days prior to randomization or anticipation of the need for major surgery during the course of study treatment
* Current peripheral neuropathy Grade >/= 2 per National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI CTCAE, v4.0)
* History of systemic anti-cancer therapy after the diagnosis of metastatic breast cancer (MBC) or for recurrent locally advanced disease, with the exception of prior hormonal regimens for recurrent locally advanced disease or MBC
* An interval of < 12 months after the last dose of vinca alkaloid or taxane chemotherapy (i.e., for treatment of early stage, non-metastatic disease)
* Hormonal therapy < 7 days prior to randomization
* Trastuzumab < 21 days prior to randomization
* Lapatinib </= 14 days prior to randomization
* Prior trastuzumab emtansine therapy
* Treatment with any other anti-cancer therapy/investigational drug (not defined above) within 21 days prior to randomization
* History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other malignancies with an expected curative outcome
* Current chronic daily treatment with corticosteroids (dose > 10 mg/day methylprednisone equivalent)
* History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab, murine proteins, docetaxel or paclitaxel
* Known hypersensitivity any of the study drugs, including excipients, or any drugs formulated in polysorbate 80

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Sabah, Sabah, Malaysia
- South Korea (3):
  - Daegu
  - Gyeonggi-do
  - Seoul
- Taiwan (2):
  - Taipei
  - Taoyuan District
- Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only 49 participants of the originally planned 561 participants were enrolled in the study at the time of study termination.
Groups:
- Arm A: Trastuzumab Emtansine: Participants were administered trastuzumab emtansine once every three weeks (Q3W). Participants could remain on study treatment until investigator assessed disease progression, unacceptable toxicity, or Sponsor study termination occurs, whichever occurs first.
  Trastuzumab Emtansine: Trastuzumab emtansine 3.6 milligrams/kilogram (mg/kg) was administered intravenously (IV) over 30-90 minutes Q3W.
- Arm B: Trastuzumab + Docetaxel: Participants were administered trastuzumab plus docetaxel Q3W. Participants could remain on study treatment until investigator assessed disease progression, unacceptable toxicity, or Sponsor study termination occurs, whichever occurs first.
  Trastuzumab: For the first three-week cycle, trastuzumab was administered IV at 8 mg/kg. For subsequent cycles, trastuzumab was administered IV at 6 mg/kg Q3W.
  Docetaxel: Docetaxel was administered IV at either 75 milligrams/square meter (mg/m^2) or 100 mg/m^2 Q3W.
Period: Overall Study
Arm/Group | Arm A: Trastuzumab Emtansine | Arm B: Trastuzumab + Docetaxel
Started | 34 | 15
Completed | 0 | 0
Not Completed | 34 | 15
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 11 | 3
Not completed — Study Terminated by Sponsor | 18 | 12
Not completed — Other | 3 | 0

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population included all randomized participants grouped according to the treatment assigned at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Trastuzumab Emtansine | Arm B: Trastuzumab + Docetaxel | Total
Number analyzed (Participants) | 34 | 15 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (9.5) | 51.7 (11.1) | 53.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 15 | 49
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from randomization to the first occurrence of disease progression or death from any cause, whichever occurred first, on the basis of investigator assessments. Progression was defined according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as at least a 20% increase in the sum of diameters of target lesions with an absolute increase of at least 5 millimeter (mm) or the appearance of one or more new lesions.
Time Frame: At time of clinical data cut-off (up to 20 months)
Population: The intent-to-treat (ITT) population included all randomized participants grouped according to the treatment assigned at randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Trastuzumab Emtansine | Arm B: Trastuzumab + Docetaxel
Number analyzed (Participants) | 34 | 15
months | 10.3 [4.2 to NA] — Not Available (NA) = parameter not estimable due to small number of participants included in analysis | 8.2 [6.0 to 13.8]

2. Primary Outcome: Safety: Percentage of Participants With Adverse Events (AEs)
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: At time of clinical data cut-off (up to 20 months)
Population: The safety analysis population consisted of all participants who received at least one dose of study drug. Safety analyses were based on the treatment that participants actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Trastuzumab Emtansine | Arm B: Trastuzumab + Docetaxel
Number analyzed (Participants) | 34 | 15
percentage of participants | 94.1 | 100

3. Primary Outcome: Safety: Percentage of Participants With Grade 3 and 4 AEs
Description: Grade 3 and 4 AEs were evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0. Grade 3 was defined as severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living, including bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden. Grade 4 was defined as life-threatening consequences; urgent intervention indicated.
Time Frame: At time of clinical data cut-off (up to 20 months)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Trastuzumab Emtansine | Arm B: Trastuzumab + Docetaxel
Number analyzed (Participants) | 34 | 15
percentage of participants | 20.6 | 66.7

4. Primary Outcome: Percentage of Participants With Adverse Events Leading to Treatment Discontinuation
Time Frame: At time of clinical data cut-off (up to 20 months)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Trastuzumab Emtansine | Arm B: Trastuzumab + Docetaxel
Number analyzed (Participants) | 34 | 15
percentage of participants | 14.7 | 20.0

5. Primary Outcome: Safety: Percentage of Participants With Adverse Events Leading to Treatment Interruption
Time Frame: At time of clinical data cut-off (up to 20 months)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Trastuzumab Emtansine | Arm B: Trastuzumab + Docetaxel
Number analyzed (Participants) | 34 | 15
percentage of participants | 11.8 | 33.3

6. Primary Outcome: Safety: Percentage of Participants With Adverse Events Leading to Dose Reduction
Time Frame: At time of clinical data cut-off (up to 20 months)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Trastuzumab Emtansine | Arm B: Trastuzumab + Docetaxel
Number analyzed (Participants) | 34 | 15
percentage of participants | 2.9 | 26.7

7. Primary Outcome: Safety: Percentage of Participants With Significant Decline in Left Ventricular Ejection Fraction (LVEF)
Description: Significant decline in LVEF was defined as LVEF below 50% and decrease from baseline of 15% points or more. Echocardiogram or multiple-gated acquisition (MUGA) scan was used to assess LVEF.
Time Frame: At time of clinical data cut-off (up to 20 months)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Trastuzumab Emtansine | Arm B: Trastuzumab + Docetaxel
Number analyzed (Participants) | 34 | 15
percentage of participants | 0 | 0

8. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause.
Time Frame: At time of clinical data cut-off (up to 20 months)
Population: The ITT population included all randomized participants grouped according to the treatment assigned at randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Trastuzumab Emtansine | Arm B: Trastuzumab + Docetaxel
Number analyzed (Participants) | 34 | 15
months | NA [NA to NA] — NA = parameter not estimable due to small number of participants included in analysis | NA [NA to NA] — NA = parameter not estimable due to small number of participants included in analysis

9. Secondary Outcome: One-Year Survival Rate
Description: One-year survival rate as determined by Kaplan-Meier estimates.
Time Frame: At 12 months
Population: The ITT population included all randomized participants grouped according to the treatment assigned at randomization. Participants, for whom data were collected, are included in the analysis for this outcome measure.
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Trastuzumab Emtansine | Arm B: Trastuzumab + Docetaxel
Number analyzed (Participants) | 8 | 8
percentage of participants | 92.31 [56.64 to 98.88] | 100.00 [NA to NA] — NA = parameter not estimable due to small number of participants included in analysis

10. Secondary Outcome: OS Truncated at 2 Years
Description: OS truncated at 2 years was defined as the time from the date of randomization to the date of death from any cause, with deaths occurring beyond 2 years after the participant's randomization date censored at 2 years.
Time Frame: At 24 months
Population: Data for this outcome measure were not collected and are therefore not reported. The study was terminated before the time point for data collection of this outcome measure.
Arm/Group | Arm A: Trastuzumab Emtansine | Arm B: Trastuzumab + Docetaxel
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as percentage of participants with partial response (PR) or complete response (CR) determined on the basis of investigator assessments with the use of RECIST v1.1. Tumor assessments were performed with computed tomography (CT) or magnetic resonance imaging (MRI) scans of the chest, abdomen, and pelvis. CR: disappearance of all target lesions; PR: >=30% decrease in the sum of the longest diameter of target lesions; Objective Response Rate (OR) = CR + PR.
Time Frame: At time of clinical data cut-off (up to 20 months)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Trastuzumab Emtansine | Arm B: Trastuzumab + Docetaxel
Number analyzed (Participants) | 27 | 14
percentage of participants | 48.1 [28.67 to 68.05] | 71.4 [41.90 to 89.60]

12. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the date of initial confirmed PR or CR to the date of disease progression or death within the study. CR: disappearance of all target lesions; PR: >=30% decrease in the sum of the longest diameter of target lesions. Disease progression was defined according to RECIST, v1.1 as at least a 20% increase in the sum of diameters of target lesions with an absolute increase of at least 5 mm or the appearance of one or more new lesions.
Time Frame: At time of clinical data cut-off (up to 20 months)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Trastuzumab Emtansine | Arm B: Trastuzumab + Docetaxel
Number analyzed (Participants) | 13 | 10
months | NA [3.5 to NA] — NA = parameter not estimable due to small number of participants included in analysis | 6.2 [4.1 to 11.7]

13. Secondary Outcome: Pharmacokinetics: Serum Concentrations of Study Medications
Description: Pharmacokinetic (PK) parameters were to be determined in a subset of participants. PK samples from the first 100 Chinese participants were planned to be collected.
Time Frame: Day 1, Cycle 1 (Day 1), Day 1, Cycle 2 (Day 22), Day 1, Cycle 4 (Day 64) and at study drug completion or discontinuation visit (up to 20 months)
Population: No PK analyses were performed as no participants were enrolled from China and no samples were collected.
Arm/Group | Arm A: Trastuzumab Emtansine | Arm B: Trastuzumab + Docetaxel
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Immunogenicity: Percentage of Positive Anti-Therapeutic Antibody (ATA) Response to Trastuzumab Emtansine
Time Frame: Day 1, Cycle 1 (Day 1), Day 1, Cycle 4 (Day 64) and at study drug completion or discontinuation visit (up to 20 months)
Population: The ITT population included all randomized participants grouped according to the treatment assigned at randomization. Only participants with at least one post-dose sample available for ATA analysis were analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Trastuzumab Emtansine
Number analyzed (Participants) | 33
percentage of participants | 3.0

15. Secondary Outcome: Patient-Reported Outcomes: Number of Participants Who Completed the Functional Assessment of Cancer Therapy-Breast Cancer (FACT-B) Questionnaire
Description: The FACT-B (version 4) is a self-reported instrument which measures health-related quality of life (HRQOL) of participants with breast cancer.The FACT-B includes the breast cancer sub-scale (BCS) and is comprised of nine items specific to assessing patients' HRQOL in breast cancer.
Time Frame: On the first Day of each 21-day Cycle (Day 1, 22, 43, etc.) and at study drug completion or discontinuation visit (up to 20 months)
Population: The ITT population included all randomized participants grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Trastuzumab Emtansine | Arm B: Trastuzumab + Docetaxel
Number analyzed (Participants) | 34 | 15
Participants
  Cycle 1 Day 1 | 34 | 15
  Cycle 2 Day 1 | 34 | 15
  Cycle 3 Day 1: number analyzed (Participants) | 33 | 15
  Cycle 3 Day 1 | 33 | 15
  Cycle 4 Day 1: number analyzed (Participants) | 30 | 14
  Cycle 4 Day 1 | 30 | 14
  Cycle 5 Day 1: number analyzed (Participants) | 27 | 13
  Cycle 5 Day 1 | 27 | 13
  Cycle 6 Day 1: number analyzed (Participants) | 23 | 12
  Cycle 6 Day 1 | 23 | 12
  Cycle 7 Day 1: number analyzed (Participants) | 18 | 11
  Cycle 7 Day 1 | 18 | 11
  Cycle 8 Day 1: number analyzed (Participants) | 16 | 11
  Cycle 8 Day 1 | 16 | 11
  Cycle 9 Day 1: number analyzed (Participants) | 15 | 10
  Cycle 9 Day 1 | 15 | 10
  Cycle 10 Day 1: number analyzed (Participants) | 12 | 7
  Cycle 10 Day 1 | 12 | 7
  Cycle 11 Day 1: number analyzed (Participants) | 11 | 7
  Cycle 11 Day 1 | 11 | 7
  Cycle 12 Day 1: number analyzed (Participants) | 9 | 7
  Cycle 12 Day 1 | 9 | 7
  Cycle 13 Day 1: number analyzed (Participants) | 8 | 5
  Cycle 13 Day 1 | 8 | 5
  Cycle 14 Day 1: number analyzed (Participants) | 7 | 5
  Cycle 14 Day 1 | 7 | 5
  Cycle 15 Day 1: number analyzed (Participants) | 6 | 4
  Cycle 15 Day 1 | 6 | 4
  Cycle 16 Day 1: number analyzed (Participants) | 3 | 4
  Cycle 16 Day 1 | 3 | 4
  Cycle 17 Day 1: number analyzed (Participants) | 2 | 2
  Cycle 17 Day 1 | 2 | 2
  Cycle 18 Day 1: number analyzed (Participants) | 2 | 1
  Cycle 18 Day 1 | 2 | 1
  Cycle 19 Day 1: number analyzed (Participants) | 1 | 1
  Cycle 19 Day 1 | 1 | 1
  Cycle 20 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 20 Day 1 | 0 | 1
  Study Drug Completion/Discontinuation Visit | 33 | 13

16. Secondary Outcome: Patient-Reported Outcomes: Number of Participants Who Completed the FACT-Taxane Questionnaire
Description: The FACT - Taxane is a self-reported instrument which measures the HRQOL of participants receiving taxane containing chemotherapy. The FACT-Taxane consists of 16 items and was designed to assess the impact of taxane treatment-related symptoms from the participant's perspective.
Time Frame: Days 1 and 8 of Cycles 1 and 2 and on the first day of each subsequent 21-day cycle thereafter as well as at study drug completion or discontinuation visit (up to 20 months)
Population: The ITT population included all randomized participants grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Trastuzumab Emtansine | Arm B: Trastuzumab + Docetaxel
Number analyzed (Participants) | 34 | 15
Participants
  Cycle 1 Day 1 | 27 | 14
  Cycle 1 Day 8 | 27 | 15
  Cycle 2 Day 1 | 29 | 15
  Cycle 2 Day 8 | 29 | 15
  Cycle 3 Day 1: number analyzed (Participants) | 33 | 15
  Cycle 3 Day 1 | 33 | 15
  Cycle 4 Day 1: number analyzed (Participants) | 30 | 14
  Cycle 4 Day 1 | 30 | 14
  Cycle 5 Day 1: number analyzed (Participants) | 27 | 13
  Cycle 5 Day 1 | 27 | 13
  Cycle 6 Day 1: number analyzed (Participants) | 23 | 12
  Cycle 6 Day 1 | 23 | 12
  Cycle 7 Day 1: number analyzed (Participants) | 18 | 11
  Cycle 7 Day 1 | 18 | 11
  Cycle 8 Day 1: number analyzed (Participants) | 16 | 11
  Cycle 8 Day 1 | 16 | 11
  Cycle 9 Day 1: number analyzed (Participants) | 15 | 10
  Cycle 9 Day 1 | 15 | 10
  Cycle 10 Day 1: number analyzed (Participants) | 12 | 7
  Cycle 10 Day 1 | 12 | 7
  Cycle 11 Day 1: number analyzed (Participants) | 11 | 7
  Cycle 11 Day 1 | 11 | 7
  Cycle 12 Day 1: number analyzed (Participants) | 9 | 7
  Cycle 12 Day 1 | 9 | 7
  Cycle 13 Day 1: number analyzed (Participants) | 8 | 5
  Cycle 13 Day 1 | 8 | 5
  Cycle 14 Day 1: number analyzed (Participants) | 7 | 5
  Cycle 14 Day 1 | 7 | 5
  Cycle 15 Day 1: number analyzed (Participants) | 6 | 4
  Cycle 15 Day 1 | 6 | 4
  Cycle 16 Day 1: number analyzed (Participants) | 3 | 4
  Cycle 16 Day 1 | 3 | 4
  Cycle 17 Day 1: number analyzed (Participants) | 2 | 2
  Cycle 17 Day 1 | 2 | 2
  Cycle 18 Day 1: number analyzed (Participants) | 2 | 1
  Cycle 18 Day 1 | 2 | 1
  Cycle 19 Day 1: number analyzed (Participants) | 1 | 1
  Cycle 19 Day 1 | 1 | 1
  Cycle 20 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 20 Day 1 | 0 | 1
  Study Drug Completion/Discontinuation Visit | 33 | 13

ADVERSE EVENTS:
Time Frame: Up to 19 months
Description: The safety analysis population consisted of all participants who received at least one dose of study drug. Safety analyses were based on the treatment that participants actually received.
Arm/Group | Arm A: Trastuzumab Emtansine | Arm B: Trastuzumab + Docetaxel
Serious Adverse Events (participants affected / at risk) | 8/34 | 5/15
Other Adverse Events (participants affected / at risk) | 31/34 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Trastuzumab Emtansine (N=34) | Arm B: Trastuzumab + Docetaxel (N=15)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Pneumonia (Infections and infestations) | 2 | 1
Post procedural cellulitis (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Trastuzumab Emtansine (N=34) | Arm B: Trastuzumab + Docetaxel (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 1
Lacrimation decreased (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4
Constipation (Gastrointestinal disorders) | 1 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 11
Dry mouth (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 11 | 3
Stomatitis (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 5
Asthenia (General disorders) | 4 | 1
Catheter site pain (General disorders) | 0 | 1
Chest discomfort (General disorders) | 2 | 0
Chills (General disorders) | 3 | 0
Device occlusion (General disorders) | 0 | 1
Extravasation (General disorders) | 1 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 9 | 1
Feeling cold (General disorders) | 3 | 1
Generalised oedema (General disorders) | 0 | 4
Malaise (General disorders) | 0 | 2
Mucosal inflammation (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 2 | 5
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 3 | 3
Central nervous system infection (Infections and infestations) | 0 | 1
Groin infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 2
Laryngitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 13 | 4
Urinary tract infection (Infections and infestations) | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 6 | 0
Aspartate aminotransferase increased (Investigations) | 8 | 1
Blood cholesterol increased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 3 | 0
Weight increased (Investigations) | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 6 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Dizziness (Nervous system disorders) | 3 | 4
Headache (Nervous system disorders) | 11 | 5
Hypoaesthesia (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 2
Paraesthesia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 8
Hallucination, auditory (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 3
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Breast discharge (Reproductive system and breast disorders) | 2 | 0
Breast pain (Reproductive system and breast disorders) | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 10
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 3
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 3 | 1

LIMITATIONS AND CAVEATS:
Due to early termination of the study only limited data from a small subset (49) of the originally planned study population size (561) are available and were too limited to perform originally planned efficacy analyses as specified in the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.